CLINICAL TRIAL: NCT04287335
Title: Stool KRAS Mutation, BMP3/NDRG4 Methylation and FIT Panel Test for the Detection of Colorectal Advanced Neoplasia in High Risk Chinese Patients
Brief Title: Multitarget Stool FIT-DNA Study for Colorectal Cancer Early Screening in China
Acronym: CLEAR-C
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: New Horizon Health Technology Co., Ltd (Unknown); Beijing Mingze Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Ding Ke-Feng, Chief physician, Zhejiang University
Other Study IDs: CLEAR-C 2018
Record Dates: First submitted 2020-02-20; First posted 2020-02-27 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Cancer; Adenomatous Polyps; Adenoma; Advanced Adenoma
Keywords: Cancer; Colorectal Cancer; Colorectal Neoplasms; Adenomatous Polyps; Adenoma; Advanced adenoma; Gastrointestinal Diseases; Colonic Diseases; Neoplasms; Digestive System Diseases; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Intestinal Diseases; Rectal Diseases; Glandular and Epithelial; Neoplasms by Histologic Type
MeSH Terms: conditions — Colorectal Neoplasms; Adenomatous Polyps; Adenoma; Neoplasms; Gastrointestinal Diseases; Colonic Diseases; Digestive System Diseases; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Intestinal Diseases; Rectal Diseases; Neoplasms by Histologic Type | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High risk CRC screening group: Prospective enrollment of subjects with pre-defined high risk factors for developing colorectal cancer
  Interventions: Diagnostic Test: Multitarget stool FIT-DNA test - ColoClear; Diagnostic Test: FIT; Procedure: Colonoscopy
- CRC group: Retrospective enrollment of subjects with confirmed colorectal cancer
  Interventions: Diagnostic Test: Multitarget stool FIT-DNA test - ColoClear; Diagnostic Test: FIT; Procedure: Colonoscopy

INTERVENTIONS:
Diagnostic Test: Multitarget stool FIT-DNA test - ColoClear — Multitarget stool FIT-DNA test
Diagnostic Test: FIT — fecal immunochemical test
Procedure: Colonoscopy — diagnostic colonoscopy

SUMMARY:
The primary objective is to determine the diagnostic sensitivity and specificity of the newly developed multitarget FIT-DNA Colorectal Cancer (CRC) screening test (ColoClear) for detecting advanced neoplasia (including colorectal cancer and advanced adenomas) in high risk patients, using colonoscopy as the reference method. The secondary objective is to compare the screening performance of the multitarget FIT-DNA test with commercially available FIT (Fecal Immunochemical Test) assay in detecting advanced neoplasia.

DETAILED DESCRIPTION:
The study will be carried out in 8 tier-3A hospitals throughout China. Patients who are at high risk of developing colorectal cancer and willing to conduct colonoscopy examination will be asked to collect stool sample prior to bowl preparation for multitarget FIT-DNA test and commercially available FIT assay. Colonoscopy and histopathologic examination are used as reference.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written consent
* Able to provide stool sample

For high risk CRC screening group:

* Scheduled for colonoscopy voluntarily or by physician prescription
* CRC high risk profile as defined below:
* History of FIT positivity
* Family history of CRC
* Any of two of the following clinical symptoms: chronic constipation/diarrhea, stool with mucous, chronic appendicitis, chronic bilary track diseases, mental stress

For CRC group:

* Confirmed CRC patients
* No prior treatment with chemotherapy, radiotherapy, and prior to any surgical procedures

Exclusion Criteria:

* Unwilling to provide stool samples
* FAP (familial adenomatous polyposis), Crohn's disease, ulcerative colitis
* Prior history of colonoscopy within the past 5 years and removal of lesions
* History of CRC
* other conditions deemed not suited for the study by investigators

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with high risk of developing CRC and patients with confirmed CRC
Sampling Method: Non-Probability Sample
Enrollment: 4758 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-12-08 (Actual); Study Completion 2020-09-13 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the ColoClear screening test with comparison to colonoscopy | Through study completion, an average of 1 year
  A diagnostic colonoscopy procedure is the reference method. Lesions will be confirmed as malignant by histopathologic examination. The DNA test includes molecular assays for KRAS mutations, aberrant NDRG4 and BMP3 methylation, plus a hemoglobin immunoassay. A logistic-regression algorithm incorporating all the above parameters was deployed to compute a single composite score, with values of 165 or more considered to be positive. The tests were processed independently of colonoscopy procedure.

SECONDARY OUTCOMES:
Sensitivity of the ColoClear screening test with comparison to FIT, with respect to advanced adenoma (AA) and CRC | Through study completion, an average of 1 year
  A diagnostic colonoscopy procedure is the reference method. Lesions will be confirmed as malignant by histopathologic examination. The ColoClear and FIT test were performed on the same stool sample.

CONTACTS AND LOCATIONS:
Overall Officials: Kefeng Ding, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (8):
- China (8):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No